CLINICAL TRIAL: NCT02605460
Title: Chemo Sensitization Before Hematopoietic Stem Cell Transplantation With a CXCR4 Antagonist in Patients With Acute Leukemia in Complete Remission: Pilot Study
Brief Title: Chemo Sensitization Before Hematopoietic Stem Cell Transplantation in Patients With Acute Leukemia in Complete Remission
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCMNSZ REF 917
Record Dates: First submitted 2015-11-09; First posted 2015-11-16 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoid Leukemia
Keywords: Bone Marrow Transplantation; Conditioning Regimen
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Busulfan; Cyclophosphamide; plerixafor; Hematopoietic Stem Cell Transplantation; Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Unique (Other): Patients will receive reduced Busulfan and Cyclophosphamide (BUCY) 2 conditioning regimen, consisting in the administration of two medications: Busulfan and Cyclophosphamide Plus: CXCR4 Antagonist. Then they will undergo a Hematopoietic Stem Cell Transplantation (Autologous or Allogeneic)
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: CXCR4 Antagonist; Procedure: Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Drug: Busulfan — 12mg/kg, Oral, divided in 4 days, 3mg/kg/day Oral, during days -7, -6, -5 y -4.
  Other Names: Myleran
Drug: Cyclophosphamide — 80mg/kg, Intravenous (IV), divided in 2 days, 40mg/kg/day IV, during days -3 y -2.
  Other Names: Cytoxan
Drug: CXCR4 Antagonist — 24mg, Subcutaneous (SC), in one day, 24mg/day SC, during day -4.
  Other Names: Plerixafor; Mozobil
Procedure: Hematopoietic Stem Cell Transplantation — Peripheral blood HSC (autologous HSCT) or Bone Marrow HSC (allogeneic HSCT) transfusion, day 0
  Other Names: Bone Marrow Transplantation

SUMMARY:
The purpose of this study is to evaluate the disease free survival and the overall survival in patients with acute leukemia in first or second complete remission after administrating a CXCR4 antagonist, as a chemo sensitization strategy, plus chemotherapy as the conditioning regimen for autologous or allogeneic hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
In the last decade, HSCT has become an efficient strategy for the treatment of many malignant and non-malignant hematological diseases, being the most common, according to the European Bone Marrow Transplantation (EBMT), acute leukemias. Both myeloid and lymphoid acute leukemias are considered malignant clonal diseases of the hematopoietic stem cells, and represent a therapeutic challenge due to the high relapse rate and mortality using conventional chemotherapy regimens. HSC reside mainly within the bone marrow, protected by a microenvironment or niche, which is perivascular, created partly by mesenchymal stromal cells and endothelial cells. Interactions between these cells and many adhesion molecules are considered a key factor for growing, transformation, and migration of neoplastic cells. The main pathway involved in the cellular transit regulation is chemokine receptor 4 (CXCR4) and its chemokine ligand 12 (CXCL12), responsible of mediating interactions between the HSC and stromal cells, and whose blocking through other cytokines and antagonists of the CXCR4 receptor (plerixafor) favors chemotaxis and HSC output to peripheral blood. Such strategy has become an effective technique to increase mobilization and harvesting in patients undergoing stem cell transplantations.

On the other hand, some preclinical studies have shown that the activation of CXCL12 pathway favors tumor growth, promoting survival and invasion of the malignant cells, recruiting stromal cells that facilitate their proliferation and promote angiogenesis directly. In such way, this pathway has been considered a therapeutic target to block their activity and inhibit tumor progression.

Patients with acute leukemia in first or second complete remission undergoing autologous or allogeneic hematopoietic stem cell transplantation (HSCT), commonly present low response rates and low survival due to persistent minimal residual disease, despite conventional high dose chemotherapy regimens. It is necessary to create strategies to increase the destruction rate of neoplastic cells in patients with acute leukemia candidates to HSCT. Our hypothesis is that the administration of a CXCR4 antagonist as part of the conditioning regimen in patients with acute leukemia candidates to HSCT will allow the mobilization and sensitization of leukemia blast cells, eradicating efficiently the minimal residual disease, responsible of posterior relapse, and will achieve a higher response rate and survival of patients undergoing this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL), candidates to HSCT
* Allogeneic HSCT: High risk AML in first complete remission (CR), AML in second CR, and ALL in first or second CR with a matched or half-matched (haploidentical) related or unrelated donor
* Autologous HSCT: Intermediate risk AML in first CR, ALL in first or second CR without a donor
* Normal liver function enzyme tests
* Preserved renal function
* Eastern Cooperative Oncology Group score ≤2 or Karnofsky ≥80%
* Left ventricle ejection fraction (LVEF) >40%
* Hemoglobin (Hb) ≥ 10 g/dl, Absolute Neutrophil Count ≥ 1 x 103/mm3, and Platelets ≥ 100,000 /µL
* Signed Informed Consent

Exclusion Criteria:

* Patients not willing to participate or to sign the informed consent
* Patients who do not meet the inclusion criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | One year
  Time from HSCT to death from any cause.

SECONDARY OUTCOMES:
Disease Free Survival | One year
  Time from HSCT to relapse of the underlying disease.

CONTACTS AND LOCATIONS:
Overall Officials: Eucario Leon Rodriguez, M.D., Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Monica M Rivera Franco, M.D.,MSc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Jantunen E. Novel strategies for blood stem cell mobilization: special focus on plerixafor. Expert Opin Biol Ther. 2011 Sep;11(9):1241-8. doi: 10.1517/14712598.2011.601737. PMID 21806478
- [Background] DiPersio JF, Ho AD, Hanrahan J, Hsu FJ, Fruehauf S. Relevance and clinical implications of tumor cell mobilization in the autologous transplant setting. Biol Blood Marrow Transplant. 2011 Jul;17(7):943-55. doi: 10.1016/j.bbmt.2010.10.018. Epub 2010 Oct 22. PMID 20971201
- [Background] Duda DG, Kozin SV, Kirkpatrick ND, Xu L, Fukumura D, Jain RK. CXCL12 (SDF1alpha)-CXCR4/CXCR7 pathway inhibition: an emerging sensitizer for anticancer therapies? Clin Cancer Res. 2011 Apr 15;17(8):2074-80. doi: 10.1158/1078-0432.CCR-10-2636. Epub 2011 Feb 24. PMID 21349998
- [Background] Redjal N, Chan JA, Segal RA, Kung AL. CXCR4 inhibition synergizes with cytotoxic chemotherapy in gliomas. Clin Cancer Res. 2006 Nov 15;12(22):6765-71. doi: 10.1158/1078-0432.CCR-06-1372. PMID 17121897
- [Background] Nervi B, Ramirez P, Rettig MP, Uy GL, Holt MS, Ritchey JK, Prior JL, Piwnica-Worms D, Bridger G, Ley TJ, DiPersio JF. Chemosensitization of acute myeloid leukemia (AML) following mobilization by the CXCR4 antagonist AMD3100. Blood. 2009 Jun 11;113(24):6206-14. doi: 10.1182/blood-2008-06-162123. Epub 2008 Dec 2. PMID 19050309
- [Background] Uy GL, Rettig MP, Motabi IH, McFarland K, Trinkaus KM, Hladnik LM, Kulkarni S, Abboud CN, Cashen AF, Stockerl-Goldstein KE, Vij R, Westervelt P, DiPersio JF. A phase 1/2 study of chemosensitization with the CXCR4 antagonist plerixafor in relapsed or refractory acute myeloid leukemia. Blood. 2012 Apr 26;119(17):3917-24. doi: 10.1182/blood-2011-10-383406. Epub 2012 Feb 2. PMID 22308295